CLINICAL TRIAL: NCT02730910
Title: Bioavailability of Anthocyanins and Phenolic Acids and Changes in Blood Antioxidant Capacity After Consumption of Purple Wheat Anthocyanin-enriched Crackers and Granola Bars by Healthy Adult Participants
Brief Title: Anthocyanin & Phenolic Acids Bioavailability & Antioxidant Capacity After Consumption of Purple Wheat Products in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Amanda Wright, Ph.D., Associate Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UGuelph
Record Dates: First submitted 2016-01-21; First posted 2016-04-07 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: Bioavailability; adults

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purple Wheat Crackers (Experimental): Bran-enriched purple wheat wholegrain crackers served in 120 g portion.
  Interventions: Other: Purple Wheat Crackers
- Purple Wheat Granola Bars (Experimental): Bran-enriched purple wheat wholegrain granola bars served in 160 g portion.
  Interventions: Other: Purple Wheat Granola Bars

INTERVENTIONS:
Other: Purple Wheat Crackers — Whole grain crackers manufactured with purple wheat
  Arms: Purple Wheat Crackers
Other: Purple Wheat Granola Bars — Whole grain granola bars manufactured with purple wheat
  Arms: Purple Wheat Granola Bars

SUMMARY:
This study will determine the bioavailability of anthocyanins and phenolic compounds from two purple wheat products, i.e. bran-enriched wholegrain purple wheat crackers and bran-enriched wholegrain purple wheat granola bars. Crackers are an example of a baked/ processed product. The purple wheat granola bars are an example of a food product that requires much less intensive preparation and cooking, compared to the crackers. A comparison of bioavailability between these two products should provide insights about how different processes and food matrix influence anthocyanin bioavailability and metabolism.

DETAILED DESCRIPTION:
This study will determine the bioavailability of anthocyanins and phenolic compounds from two purple wheat products, i.e. bran-enriched wholegrain purple wheat crackers and bran-enriched wholegrain purple wheat granola bars. Crackers are an example of a baked/ processed product. The purple wheat granola bars are an example of a food product that requires much less intensive preparation and cooking, compared to the crackers. A comparison of bioavailability between these two products should provide insights about how different processes and food matrix influence anthocyanin bioavailability and metabolism. The study is a crossover investigation with 8 men and 8 women who will adhere to a low anthocyanin and low phenolic diet for the duration and complete 2 postprandial study visits where, in random order, they will consume either the crackers or granola bars. Blood and urine will be collected at baseline and postprandially for the analysis of anthocyanins and their metabolites and phenolic acids and determination of antioxidant capacity.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18 - 27 kg/m2
* Generally healthy as determined by screening questionnaire
* Non-smoking
* Non to moderate alcohol drinkers (Typical consumption less than 5 drinks per sitting and no more than 14 per week)

Exclusion Criteria:

* Pregnant or breast-feeding females
* History of any major disease or medical condition, including any disorder of the gastrointestinal system or food intolerances
* Taking any prescription medications (including hormonal contraceptives) or over the counter medications prescribed by a medical professional
* Taking any natural health products or dietary supplements, other than a multivitamin low in anthocyanins and phenolic acids
* Oral antibiotic use in the past 3 months
* Any food allergies, and any anaphylactic or life-threatening allergies - food or otherwise
* Smokers or use of recreational drugs (marijuana, magic mushrooms, etc)
* Elite or training athletes
* Following a vegan or vegetarian diet

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of anthocyanin metabolites | 0-8 hours (0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8)

SECONDARY OUTCOMES:
Plasma concentrations of phenolic acids | 0-8 hours (0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8)
Plasma antioxidant capacity | 0-8 hours (0, 2, 4, 6, 8)
Urinary concentrations of phenolic acids | 0-8 hours (0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8)
Urinary concentrations of anthocyanin metabolites | 0-8 hours (0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutraceutical Research Unit, University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Through peer reviewed publications